CLINICAL TRIAL: NCT03354819
Title: Effects of a Modified Mindfulness-based Cognitive Therapy for Family Caregivers of People With Dementia in Stress Reduction: A Randomized Controlled Trial
Brief Title: Effects of a Modified Mindfulness-based Cognitive Therapy for Family Caregivers of People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Patrick KOR Pui Kin, PhD candidate, Center for Gerontological Nursing, School of Nursing, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSEARS20170929002
Record Dates: First submitted 2017-11-17; First posted 2017-11-28 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Carer Stress Syndrome; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: A prospective, single-blind, parallel-group randomized controlled trial (RCT) will be adopted to test the hypotheses and compare the immediate effects and its effects over a 3-month follow up between the MBCT program and an active control group (social interactions and routine education on dementia care) for the family caregivers of PWD in the community. The MBCT program consists of seven sessions, including different mindfulness activities (such as mindful eating and mindful walking) and peer sharing, while the parallel active control group will have the social interactions and routine education on dementia care, including seven education sessions on dementia care, caregiver skills training and group sharing, aiming to control/balance the social interaction effects that can also be found in the MBI group. The study will also follow the guideline recommended by the latest Consolidated Standards of Reporting Trials (Schulz et al., 2010) statements.
Who Masked: Outcomes Assessor
Masking Description: The eligible participants will be randomized into the 2 groups (MBCT and SIRE), following the allocation concealment mechanism by an independent assistant. The research assistants who were blinded to the group assignment performed all of the outcome measurements and data entries. The procedure and treatment allocation will be blinded to the investigator and the interventionists until the baseline measurement is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified MBCT (Experimental): A group-based, 10-week, 7-session modified Mindfulness Based Cognitive Therapy (MBCT) will be adopted in the MBCT intervention group with a group size of 15-20. The program includes different mindfulness activities (such as mindful eating and mindful walking) and peer sharing.
  Interventions: Behavioral: Modified MBCT
- SIRE on dementia (Active Comparator): The frequency of the Social Interactions and Routine Education (SIRE) program is the same as that of modified MBCT which consists of seven sessions (weekly for the first four sessions and bi-weekly for the last three sessions) and each session will last about two hours for 10 weeks with group size 15-20.
  Interventions: Behavioral: SIRE on dementia

INTERVENTIONS:
Behavioral: Modified MBCT — Compared with the original protocol of Mindfulness-based Cognitive Therapy (Segal et al., 2002), the modified MBCT protocol in this pilot study has the following changes:
  Outline:
  Session 1 Awareness and automatic pilot:
  Session 2 Living in our head
  Session 3 Gathering the scattered mind
  Session 4 Recognizing aversion & allowing
  Session 5 Thoughts are not facts
  Session 6 Take care of myself
  Session 7 Maintaining and extending new learning
  Arms: Modified MBCT
Behavioral: SIRE on dementia — The SIRE program includes routine education sessions on dementia care, caregiver skills training, and group sharing on caregiving tasks.
  Outline:
  1. Overview of dementia
  2. Pharmacological and non-pharmacological treatment of dementia
  3. BPSD in dementia care
  4. Person center care
  5. Advance planning in people with dementia
  6. Principle of mindfulness
  7. Non-pharmacological intervention on stress reduction
  Arms: SIRE on dementia

SUMMARY:
Caring for people with dementia (PWD) poses many challenges which may cause high levels of caregiver stress. This study aims to investigate the effects of a modified Mindfulness-based Cognitive Therapy for stress reduction in the family caregivers of PWD. A prospective, single-blind, parallel-group randomized controlled trial (RCT) of 76 family caregivers of PWD will be recruited and randomized to either the MBCT or the control groups.The primary outcomes (stress) and secondary outcomes (anxiety, depression, burden, quality of life and resilience) will be measured at immediate post-intervention (T1) and at 3 months follow up (T2) which will be compared with the baseline (T0). Mixed repeated measure MANOVA will be performed to assess the effects of time, group, and time-group interaction on all outcome measurements.To understand the therapeutic components and identify the strengths, limitations, and difficulties of the MBCT program, process evaluation will be conducted through focus group interviews with 15 participants from the MBI group. It is hypothesized that the MBCT group will have a significantly greater reduction of stress (primary outcome) and improvement in the secondary outcomes, namely depression, anxiety, and burden, at T1 and/or T2 than the control group.

DETAILED DESCRIPTION:
Background:

Caring for people with dementia (PWD) poses many challenges which may cause high levels of caregiver stress. Mindfulness-based intervention (MBI) is a newly adopted psychosocial intervention through an integration of the mind and body to reduce stress of the participants. A systematic review was conducted with five studies (four RCTs and one quasi-experimental study) to investigate the effect of MBI in stress reduction in the family caregivers of PWD. Of these, three trials involving 144 participants were eligible for the meta-analysis. The result showed that the stress levels dropped significantly after an 8-week MBI in the family caregivers of PWD with a moderate aggregated effect size of 0.57 (95% CI [0.23, 0.92], overall effect Z= 3.25 at p= 0.001). While MBI's immediate effect was found, the long term effect was unclear. Besides a limited number of clinical trials and several limitations (such as poor study design and small sample size) were also identified in this review. It signifies that more studies are still required to examine the effects of MBI for family caregivers of PWD. Since MBI is a new intervention for stress management among the family caregivers of PWD, a feasibility study was conducted between 2016 and 2017. It found that the family caregivers could master the mindfulness skill after the mindfulness sessions with a low attrition rate of 3.8%. A modified Mindfulness-based cognitive therapy (MBCT) protocol was also validated in the study to fit the local need and address the limitations identified in previous studies.

Objective:

This study aims to investigate the effects of a modified MBCT for stress reduction in the family caregivers of PWD in Hong Kong.

Methods:

A prospective, single-blind, parallel-group randomized controlled trial (RCT) of 76 family caregivers of PWD will be recruited and randomized to either the MBCT or the control groups. The MBI groups will receive a seven-week, group-based MBCT training whereas the control group will receive social interactions and routine education on dementia care program of a frequency and timing similar to those of the MBI group. The primary outcomes (stress) and secondary outcomes (anxiety, depression, burden, quality of life, resilience) will be measured at immediate post-intervention (T1) and at 3 months follow up (T2) which will be compared with the baseline (T0). Mixed repeated measure MANOVA will be performed to assess the effects of time, group, and time-group interaction on all outcome measurements. Both per-protocol (PP) and intention-to-treat (ITT) analysis will be performed in order to find out more factors affecting the use and effectiveness of MBCT such as non-compliance and acceptability. To understand the therapeutic components and identify the strengths, limitations, and difficulties of the MBCT program, process evaluation will be conducted through focus group interviews with 15 participants from the MBI group. It is hypothesized that the MBCT group will have a significantly greater reduction of stress (primary outcome) and improvement in the secondary outcomes, namely anxiety, depression, burden, quality of life, and resilience at T1 and/or T2 than the control group.

Significance and Value:

Reducing the caregiving stress level can promote the well-being of the family caregivers to maintain their sustainability in terms of providing daily care for their family members with dementia for a longer period of time. Evidence shows a minimal and short term effects of other psychosocial interventions (such as respite care, mutual support group) for reducing caregivers' stress. On the other hand, the MBCT is found effective in stress reduction in other populations. This finding is also supported by a feasibility study of using the MBI in family caregivers of PWD. The results of this study may be able to provide us with evidence for using MBCT as a standard supportive intervention for the family caregivers of PWD.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or above;
2. the blood or by-marriage relatives (e.g. spouses, siblings, children, and grandchildren) of a person who has been clinically diagnosed with dementia, regardless of its types (as mentioned in the operational definitions section (p. 1) and these relatives are taking up the caring responsibilities ranging from physical aids to emotional supports, in the form of transportation, financial assistance, personal hygiene, and decision-making.;
3. providing most of the daily care and support for PWD (daily contact for at least four hours); and
4. able to speak Cantonese (for understanding about all teaching materials and instructions).

Exclusion Criteria:

1. are practicing or recently learned meditation, mindfulness activities, and/or relaxation training in the past 6 months;
2. are diagnosed with a mental disorder such as bipolar disorder, schizophrenia, dementia, or depression; and/or,
3. are taking anticonvulsants, or any kind of psychotropic drugs, and/or identified with a self-reported suicidal thought or drug abuse in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-12-23 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-06-23 (Actual)

PRIMARY OUTCOMES:
Change of Perceived Stress Scale (PSS) | At baseline (T0), 10th week (immediately post- intervention; T1), and 3 months after the intervention (follow-up assessment, T2)
  Perceived Stress Scale contains 10 items with 5-point Likert-type scale rating from 0 (never) to 4 (very often). The total score can range from 0 to 40 with higher scores indicating higher perceived stress.
  Comparisons of changes of Perceived Stress Scale will be considered as follows:
  T0 - T1; T0 - T2; T1 - T2

SECONDARY OUTCOMES:
Zarit Burden Scale (ZBI). | At baseline (T0), 10th week (immediately post- intervention; T1), and 3 months after the intervention (follow-up assessment, T2)
  Zarit Burden Scale comprises of 22 items including factors most frequently mentioned by caregivers as problem areas such as carer's health, psychological well-being, and the relationships between the carer and the patient with dementia. The score can range from 0 to 88. A higher score indicates greater carer distress.
  Comparisons of changes of Zarit Burden Scale will be considered as follows:
  T0 - T1; T0 - T2; T1 - T2
Change of Center for Epidemiologic Studies Depression Scale (CESD) | At baseline (T0), 10th week (immediately post- intervention; T1), and 3 months after the intervention (follow-up assessment, T2)
  Center for Epidemiologic Studies Depression Scale is a self-reported measure of depression containing 20 items. It measures the common symptoms of depression in term of depressed mood, feelings of guilt and worthlessness, and feelings of helplessness. The scores can range from 0 to 60 and higher CESDS scores indicate increasing levels of depression.
  Comparisons of changes of Center for Epidemiologic Studies Depression Scale will be considered as follows:
  T0 - T1; T0 - T2; T1 - T2
Change of Hospital Anxiety and Depression Scale (HADS) | At baseline (T0), 10th week (immediately post- intervention; T1), and 3 months after the intervention (follow-up assessment, T2)
  The level of anxiety will be measured by the Hospital Anxiety and Depression Scale which is a 7-item self-report instrument including specific items that assess generalized anxiety including tension, worry, fear, panic, difficulties in relaxing, and restlessness. The scores range from 0 to 21 and higher scores indicate increasing levels of anxiety
  Comparisons of changes of Hospital Anxiety and Depression Scale will be considered as follows:
  T0 - T1; T0 - T2; T1 - T2
Change of Brief Resilience Scale (BRS) | At baseline (T0), 10th week (immediately post- intervention; T1), and 3 months after the intervention (follow-up assessment, T2)
  The level of resilience (the ability to bounce back or recover from stress) will be measured by the Brief Resilience Scale, which is a 6-item, self-report and 5-point rating scale. The scores can range from 6 to 30 with higher scores indicating higher level of resilience.
  Comparisons of changes of Brief Resilience Scale will be considered as follows:
  T0 - T1; T0 - T2; T1 - T2
Change of 12-Item Short Form Health Survey | At baseline (T0), 10th week (immediately post- intervention; T1), and 3 months after the intervention (follow-up assessment, T2)
  Caregivers' health-related quality of life will be measured by 12-Item Short Form Health Survey. It contains twelve questions and ranges from 0 to 100, where a zero score indicates the lowest level of healthmeasured by the scales and 100 indicates the highest level of health
  Comparisons of changes of 12-Item Short Form Health Survey will be considered as follows:
  T0 - T1; T0 - T2; T1 - T2

OTHER OUTCOMES:
Change of Five Facets Mindfulness Questionnaire-Short Form | At baseline (T0), 10th week (immediately post- intervention; T1), and 3 months after the intervention (follow-up assessment, T2)
  Caregivers' level of mindfulness will be measured as the process indicator by using the Five Facets Mindfulness Questionnaire Short Form. It is a self-report questionnaire measuring the five facets of mindfulness which includes observing, describing, acting with awareness, non-judging of inner and non-reactivity to inner experience (e.g., "I'm good at finding words to describe my feelings"). The total score ranges from 20 to 100 and the higher the score, the higher level of mindfulness.
  Comparisons of changes of Five Facets Mindfulness Questionnaire-Short Form will be considered as follows:
  T0 - T1; T0 - T2; T1 - T2
Weekly mindfulness practice (hours) | Weekly starting from baseline T0, to 3 months after the intervention (follow-up assessment, T2)
  Weekly mindfulness practice will be measured by the average number of hours in practicing mindfulness per week from T0 to T2.
Adherence rate of intervention | Weekly starting from baseline T0 to 10th week (immediately post- intervention, T1)
  The (Number of sessions a participant is present) / (Total number of intervention sessions) will be measured to indicate the adherence rate

CONTACTS AND LOCATIONS:
Overall Officials: Justina Liu, PhD, Study Chair — The Hong Kong Polytechnic Univeristy
Locations (1):
- Patrick Kor, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adelman RD, Tmanova LL, Delgado D, Dion S, Lachs MS. Caregiver burden: a clinical review. JAMA. 2014 Mar 12;311(10):1052-60. doi: 10.1001/jama.2014.304. PMID 24618967
- [Background] Abbott RA, Whear R, Rodgers LR, Bethel A, Thompson Coon J, Kuyken W, Stein K, Dickens C. Effectiveness of mindfulness-based stress reduction and mindfulness based cognitive therapy in vascular disease: A systematic review and meta-analysis of randomised controlled trials. J Psychosom Res. 2014 May;76(5):341-51. doi: 10.1016/j.jpsychores.2014.02.012. Epub 2014 Mar 11. PMID 24745774
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Barnhofer T, Crane C, Hargus E, Amarasinghe M, Winder R, Williams JM. Mindfulness-based cognitive therapy as a treatment for chronic depression: A preliminary study. Behav Res Ther. 2009 May;47(5):366-73. doi: 10.1016/j.brat.2009.01.019. Epub 2009 Feb 5. PMID 19249017
- [Background] Bazzano, A., Wolfe, C., Zylowska, L., Wang, S., Schuster, E., Barrett, C., & Lehrer, D. (2015). Mindfulness based stress reduction (MBSR) for parents and caregivers of individuals with developmental disabilities: a community-based approach. Journal of Child and Family Studies, 24(2), 298-308. doi: 10.1007/s10826-013-9836-9
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Brown KW, Coogle CL, Wegelin J. A pilot randomized controlled trial of mindfulness-based stress reduction for caregivers of family members with dementia. Aging Ment Health. 2016 Nov;20(11):1157-1166. doi: 10.1080/13607863.2015.1065790. Epub 2015 Jul 27. PMID 26211415
- [Background] Cerejeira J, Lagarto L, Mukaetova-Ladinska EB. Behavioral and psychological symptoms of dementia. Front Neurol. 2012 May 7;3:73. doi: 10.3389/fneur.2012.00073. eCollection 2012. PMID 22586419
- [Background] Ko KT, Yip PK, Liu SI, Huang CR. Chinese version of the Zarit caregiver Burden Interview: a validation study. Am J Geriatr Psychiatry. 2008 Jun;16(6):513-8. doi: 10.1097/JGP.0b013e318167ae5b. PMID 18515696
- [Background] Chan WC, Ng C, Mok CC, Wong FL, Pang SL, Chiu HF. Lived experience of caregivers of persons with dementia in Hong Kong: a qualitative study. East Asian Arch Psychiatry. 2010 Dec;20(4):163-8. PMID 22348924
- [Background] Chan YF, Leung DY, Fong DY, Leung CM, Lee AM. Psychometric evaluation of the Hospital Anxiety and Depression Scale in a large community sample of adolescents in Hong Kong. Qual Life Res. 2010 Aug;19(6):865-73. doi: 10.1007/s11136-010-9645-1. Epub 2010 Apr 7. PMID 20373037
- [Background] Chen Y, Yang X, Wang L, Zhang X. A randomized controlled trial of the effects of brief mindfulness meditation on anxiety symptoms and systolic blood pressure in Chinese nursing students. Nurse Educ Today. 2013 Oct;33(10):1166-72. doi: 10.1016/j.nedt.2012.11.014. Epub 2012 Dec 20. PMID 23260618
- [Background] Chien, W.T., Cheung, D.S.K., Lai, C.K.Y., Yip, A.L.K., Kor, P.P.K., Moyle, W., Chambers, S., Jones, C., & Davies, N. (2017). [Use of a mindfulness-based intervention for family carers of people with dementia in the community: a feasibility study] Unpublished raw data.
- [Background] Chien WT, Thompson DR. Effects of a mindfulness-based psychoeducation programme for Chinese patients with schizophrenia: 2-year follow-up. Br J Psychiatry. 2014 Jul;205(1):52-9. doi: 10.1192/bjp.bp.113.134635. Epub 2014 May 8. PMID 24809397
- [Background] Chiesa A, Calati R, Serretti A. Does mindfulness training improve cognitive abilities? A systematic review of neuropsychological findings. Clin Psychol Rev. 2011 Apr;31(3):449-64. doi: 10.1016/j.cpr.2010.11.003. Epub 2010 Dec 1. PMID 21183265
- [Background] Chin WY, Choi EP, Chan KT, Wong CK. The Psychometric Properties of the Center for Epidemiologic Studies Depression Scale in Chinese Primary Care Patients: Factor Structure, Construct Validity, Reliability, Sensitivity and Responsiveness. PLoS One. 2015 Aug 7;10(8):e0135131. doi: 10.1371/journal.pone.0135131. eCollection 2015. PMID 26252739
- [Background] Christopher, M. S., Goerling, R. J., Rogers, B. S., Hunsinger, M., Baron, G., Bergman, A. L., & Zava, D. T. (2016). A pilot study evaluating the effectiveness of a mindfulness-based intervention on cortisol awakening response and health outcomes among law enforcement officers. Journal of Police and Criminal Psychology, 31(1), 15-28. doi:10.1007/s11896-015-9161-x
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Epstein-Lubow, G., McBee, L., Darling, E., Armey, M., & Miller, I. W. (2011). A pilot investigation of mindfulness-based stress reduction for caregivers of frail elderly. Mindfulness, 2(2), 95-102. doi: 10.1007/s12671-011-0047-4.
- [Background] Etters L, Goodall D, Harrison BE. Caregiver burden among dementia patient caregivers: a review of the literature. J Am Acad Nurse Pract. 2008 Aug;20(8):423-8. doi: 10.1111/j.1745-7599.2008.00342.x. PMID 18786017
- [Background] Fialho PP, Koenig AM, Santos MD, Barbosa MT, Caramelli P. Positive effects of a cognitive-behavioral intervention program for family caregivers of demented elderly. Arq Neuropsiquiatr. 2012 Oct;70(10):786-92. doi: 10.1590/s0004-282x2012001000007. PMID 23060105
- [Background] Garland, E., Gaylord, S., & Fredrickson, B. (2011). Positive reappraisal mediates the stress-reductive effects of mindfulness: an upward spiral process. Mindfulness, 2(1), 59-67. doi:10.1007/s12671-011-0043-8
- [Background] Gecht J, Kessel R, Forkmann T, Gauggel S, Drueke B, Scherer A, Mainz V. A mediation model of mindfulness and decentering: sequential psychological constructs or one and the same? BMC Psychol. 2014 Jul 7;2(1):18. doi: 10.1186/2050-7283-2-18. eCollection 2014. PMID 25815189
- [Background] Godfrin KA, van Heeringen C. The effects of mindfulness-based cognitive therapy on recurrence of depressive episodes, mental health and quality of life: A randomized controlled study. Behav Res Ther. 2010 Aug;48(8):738-46. doi: 10.1016/j.brat.2010.04.006. Epub 2010 Apr 18. PMID 20462570
- [Background] The Practice of Nursing Research: Appraisal, Synthesis, and Generation of Evidence - Seventh edition Grove Susan K The Practice of Nursing Research: Appraisal, Synthesis, and Generation of Evidence - Seventh edition 752pp Elsevier 9781455707362 1455707368 [Formula: see text]. Nurs Stand. 2013 Apr 3;27(31):30. doi: 10.7748/ns2013.04.27.31.30.b1488. PMID 26981669
- [Background] Hofmann SG, Asnaani A, Vonk IJ, Sawyer AT, Fang A. The Efficacy of Cognitive Behavioral Therapy: A Review of Meta-analyses. Cognit Ther Res. 2012 Oct 1;36(5):427-440. doi: 10.1007/s10608-012-9476-1. Epub 2012 Jul 31. PMID 23459093
- [Background] Holzel BK, Lazar SW, Gard T, Schuman-Olivier Z, Vago DR, Ott U. How Does Mindfulness Meditation Work? Proposing Mechanisms of Action From a Conceptual and Neural Perspective. Perspect Psychol Sci. 2011 Nov;6(6):537-59. doi: 10.1177/1745691611419671. PMID 26168376
- [Background] Hou, J. (2012) The effects of mindfulness-based stress reduction program on depressive symptoms reduction among family caregivers in Hong Kong (Doctoral dissertation) Retrieved from CUHK Electronic Theses & Dissertations Collection.
- [Background] Hou RJ, Wong SY, Yip BH, Hung AT, Lo HH, Chan PH, Lo CS, Kwok TC, Tang WK, Mak WW, Mercer SW, Ma SH. The effects of mindfulness-based stress reduction program on the mental health of family caregivers: a randomized controlled trial. Psychother Psychosom. 2014;83(1):45-53. doi: 10.1159/000353278. Epub 2013 Nov 19. PMID 24281411
- [Background] Hou J, Wong SY, Lo HH, Mak WW, Ma HS. Validation of a Chinese version of the Five Facet Mindfulness Questionnaire in Hong Kong and development of a short form. Assessment. 2014 Jun;21(3):363-71. doi: 10.1177/1073191113485121. Epub 2013 Apr 16. PMID 23596271
- [Background] Imel Z, Baldwin S, Bonus K, Maccoon D. Beyond the individual: group effects in mindfulness-based stress reduction. Psychother Res. 2008 Nov;18(6):735-42. doi: 10.1080/10503300802326038. PMID 18815948
- [Background] Jaffray L, Bridgman H, Stephens M, Skinner T. Evaluating the effects of mindfulness-based interventions for informal palliative caregivers: A systematic literature review. Palliat Med. 2016 Feb;30(2):117-31. doi: 10.1177/0269216315600331. Epub 2015 Aug 17. PMID 26281853
- [Background] Jimenez, S. S., Niles, B. L., & Park, C. L. (2010). A mindfulness model of affect regulation and depressive symptoms: Positive emotions, mood regulation expectancies, and self-acceptance as regulatory mechanisms. Personality and Individual Differences, 49(6), 645-650. doi:10.1016/j.paid.2010.05.041
- [Background] Kabat-Zinn, J. (1990). Full catastrophe living : using the wisdom of your body and mind to face stress, pain, and illness. New York:Delacorte Press.
- [Background] Kenny MA, Williams JM. Treatment-resistant depressed patients show a good response to Mindfulness-based Cognitive Therapy. Behav Res Ther. 2007 Mar;45(3):617-25. doi: 10.1016/j.brat.2006.04.008. Epub 2006 Jun 23. PMID 16797486
- [Background] Kor, P. P. K., Chien, W. T., Liu, J. Y. W., & Lai, C. K. Y. (2017) Mindfulness-based intervention for stress reduction of family caregivers of people with dementia: a systematic review and meta-analysis. Mindfulness. Advance online publication. doi: 10.1007/s12671-017-0751-9
- [Background] Lam CL, Tse EY, Gandek B. Is the standard SF-12 health survey valid and equivalent for a Chinese population? Qual Life Res. 2005 Mar;14(2):539-47. doi: 10.1007/s11136-004-0704-3. PMID 15892443
- [Background] Lam ET, Lam CL, Fong DY, Huang WW. Is the SF-12 version 2 Health Survey a valid and equivalent substitute for the SF-36 version 2 Health Survey for the Chinese? J Eval Clin Pract. 2013 Feb;19(1):200-8. doi: 10.1111/j.1365-2753.2011.01800.x. Epub 2011 Nov 29. PMID 22128754
- [Background] Lazarus, R. S., & Folkman, S. (1984). Stress, appraisal, and coping. New York: Springer
- [Background] Lebois LA, Papies EK, Gopinath K, Cabanban R, Quigley KS, Krishnamurthy V, Barrett LF, Barsalou LW. A shift in perspective: Decentering through mindful attention to imagined stressful events. Neuropsychologia. 2015 Aug;75:505-24. doi: 10.1016/j.neuropsychologia.2015.05.030. Epub 2015 Jun 22. PMID 26111487
- [Background] Leung DY, Lam TH, Chan SS. Three versions of Perceived Stress Scale: validation in a sample of Chinese cardiac patients who smoke. BMC Public Health. 2010 Aug 25;10:513. doi: 10.1186/1471-2458-10-513. PMID 20735860
- [Background] Maayan N, Soares-Weiser K, Lee H. Respite care for people with dementia and their carers. Cochrane Database Syst Rev. 2014 Jan 16;2014(1):CD004396. doi: 10.1002/14651858.CD004396.pub3. PMID 24435941
- [Background] Manicavasgar V, Parker G, Perich T. Mindfulness-based cognitive therapy vs cognitive behaviour therapy as a treatment for non-melancholic depression. J Affect Disord. 2011 Apr;130(1-2):138-44. doi: 10.1016/j.jad.2010.09.027. Epub 2010 Nov 20. PMID 21093925
- [Background] McCown, D., Reibel, D., & Micozzi, M. S. (2017). Resources for teaching mindfulness: An international handbook. New York: Springer International Publishing.
- [Background] Meinert, C. L., & Tonascia, S. (1986). Clinical trials: design, conduct, and analysis. UK: Oxford University Press
- [Background] Oken BS, Fonareva I, Haas M, Wahbeh H, Lane JB, Zajdel D, Amen A. Pilot controlled trial of mindfulness meditation and education for dementia caregivers. J Altern Complement Med. 2010 Oct;16(10):1031-8. doi: 10.1089/acm.2009.0733. Epub 2010 Oct 7. PMID 20929380
- [Background] Paller KA, Creery JD, Florczak SM, Weintraub S, Mesulam MM, Reber PJ, Kiragu J, Rooks J, Safron A, Morhardt D, O'Hara M, Gigler KL, Molony JM, Maslar M. Benefits of mindfulness training for patients with progressive cognitive decline and their caregivers. Am J Alzheimers Dis Other Demen. 2015 May;30(3):257-67. doi: 10.1177/1533317514545377. Epub 2014 Aug 25. PMID 25154985
- [Background] Radloff, L. S. (1977). The CES-D scale: A self-report depression scale for research in the general population. Applied Psychological Measurement, 1(3), 385-401. doi:10.1177/014662167700100306
- [Background] Safran, J., & Segal, Z. V. (1996). Interpersonal process in cognitive therapy. New York: Jason Aronson.
- [Background] Salzer S, Winkelbach C, Leweke F, Leibing E, Leichsenring F. Long-term effects of short-term psychodynamic psychotherapy and cognitive-behavioural therapy in generalized anxiety disorder: 12-month follow-up. Can J Psychiatry. 2011 Aug;56(8):503-8. doi: 10.1177/070674371105600809. PMID 21878162
- [Background] Santorelli, S. F. (2014). Mindfulness-based stress reduction (MBSR): Standards of practice. Retrieved from http://www.umassmed.edu/PageFiles/63144/mbsr_standards_of_practice_2014.pdf
- [Background] Schulz KF, Grimes DA. Generation of allocation sequences in randomised trials: chance, not choice. Lancet. 2002 Feb 9;359(9305):515-9. doi: 10.1016/S0140-6736(02)07683-3. PMID 11853818
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Schulz R, Martire LM. Family caregiving of persons with dementia: prevalence, health effects, and support strategies. Am J Geriatr Psychiatry. 2004 May-Jun;12(3):240-9. PMID 15126224
- [Background] Segal, Z. V., Williams, J. M. G., & Teasdale, J. D. (2002). Mindfulness-based cognitive therapy for depression : A new approach to preventing relapse. New York: Guilford Press.
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Sorensen S, Pinquart M, Duberstein P. How effective are interventions with caregivers? An updated meta-analysis. Gerontologist. 2002 Jun;42(3):356-72. doi: 10.1093/geront/42.3.356. PMID 12040138
- [Background] Speca M, Carlson LE, Goodey E, Angen M. A randomized, wait-list controlled clinical trial: the effect of a mindfulness meditation-based stress reduction program on mood and symptoms of stress in cancer outpatients. Psychosom Med. 2000 Sep-Oct;62(5):613-22. doi: 10.1097/00006842-200009000-00004. PMID 11020090
- [Background] Stratford HJ, Cooper MJ, Di Simplicio M, Blackwell SE, Holmes EA. Psychological therapy for anxiety in bipolar spectrum disorders: a systematic review. Clin Psychol Rev. 2015 Feb;35:19-34. doi: 10.1016/j.cpr.2014.11.002. Epub 2014 Nov 8. PMID 25462111
- [Background] Wang F, Feng TY, Yang S, Preter M, Zhou JN, Wang XP. Drug Therapy for Behavioral and Psychological Symptoms of Dementia. Curr Neuropharmacol. 2016;14(4):307-13. doi: 10.2174/1570159x14666151208114232. PMID 26644152
- [Derived] Kor PPK, Liu JYW, Chien WT. Effects of a Modified Mindfulness-Based Cognitive Therapy for Family Caregivers of People With Dementia: A Randomized Clinical Trial. Gerontologist. 2021 Aug 13;61(6):977-990. doi: 10.1093/geront/gnaa125. PMID 32886746
- [Derived] Kor PPK, Liu JY, Chien WT. Effects on stress reduction of a modified mindfulness-based cognitive therapy for family caregivers of those with dementia: study protocol for a randomized controlled trial. Trials. 2019 May 29;20(1):303. doi: 10.1186/s13063-019-3432-2. PMID 31142366